CLINICAL TRIAL: NCT01423162
Title: Iron Bioavailability Study Of Fortified Oat Drink
Brief Title: Iron Bioavailability of Fortified Oat Drink
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: Food and Nutrition Research Institute, Philippines (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP 1009
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-08

CONDITIONS: Iron Absorption
Keywords: Iron absorption; Oats; fortified oat beverages
MeSH Terms: interventions — Diet Therapy; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drink with Vit C then drink without Vit C (Experimental): Fortified oat drink with vitamin C on day 1 followed by fortified oat drink without vitamin C on day 2
  Interventions: Other: Dietary Intervention (with Vit C then without Vit C)
- Drink without Vit C then drink with Vit C (Experimental): Fortified oat drink without vitamin C on day 1 followed by fortified oat drink with vitamin C on day 2
  Interventions: Other: Dietary Intervention (without Vit C followed by with Vit C)

INTERVENTIONS:
Other: Dietary Intervention (with Vit C then without Vit C) — Fortified oat drink with vitamin C followed by fortified oat drink without vitamin C
  Arms: Drink with Vit C then drink without Vit C
Other: Dietary Intervention (without Vit C followed by with Vit C) — Fortified oat drink without vitamin C followed by fortified oat drink with vitamin C
  Arms: Drink without Vit C then drink with Vit C

SUMMARY:
This study will follow a double blinded randomized controlled study design to enroll 20 apparently healthy 6 year old children. The children will be fed with two different nutrient fortified oat drinks labeled with stable isotopes of iron (Fe-57 or Fe-58 as NaFeEDTA). Fourteen days after consumption of meals on Day 2, blood will be drawn from the children for stable isotope measurements and iron absorption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* 6 year old children (inclusive)
* Normal BMI for age (WHO standard: 15.3-15.5 kg)
* Apparently healthy, no metabolic or gastrointestinal disorder; non-anemic (Hemoglobin values not less than 11.5 mg/dL -WHO cut-off for respective age)
* No medication or vitamin/mineral supplement will be consumed during the study; intake of vitamin/mineral supplement will be discontinued 2 weeks before the start of the study
* Parents demonstrate an understanding of the given information and ability to comply with the study procedure
* Obtained parental or legal representative's informed consent

Exclusion Criteria:

* Known gastrointestinal or metabolic disorder or experiencing blood losses over the past 6 months;
* Children taking medication
* Children who are anemic (Hemoglobin values less than 11.5 mg/dL - WHO cut-off value for this age)
* Currently participating or having participated in another clinical trial during the past 3 months prior to the beginning of the study

Ages: 6 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trinidad P Trinidad, PhD, Principal Investigator — FNRI
Locations (1):
- Food and Nutrition Research Institute, City of Taguig, Philippines

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in August 2011
Pre-assignment Details: One subject was excluded prior to group assignment due to illness
Groups:
- Drink With Vit C Then Drink Without Vit C: Dietary Intervention: Fortified oat drink with vitamin C followed by fortified oat drink without viatamin C
- Drink Without Vitamin C Then Drink With Vit C: Dietary Intervention: Fortified oat drink without vitamin C followed by fortified oat drink with vitamin C.
Period: Overall Study
Arm/Group | Drink With Vit C Then Drink Without Vit C | Drink Without Vitamin C Then Drink With Vit C
Started | 11 | 9
Completed | 11 (Crossover design: All subjects (n=20) completed both arms) | 9 (Crossover design: All subjects (n=20) completed both arms)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Drink With Vit C Then Drink Without Vit C: Dietary Intervention (with Vitamin C): Fortified oat drink with vitamin C followed by fortified oat drink without Vit C
- Drink Without Vit C Then Drink With Vit C: Dietary Intervention (without Vitamin C): Fortified oat drink without vitamin C followed by fortified oat drink with vitamin C
- Total: Total of all reporting groups
Arm/Group | Drink With Vit C Then Drink Without Vit C | Drink Without Vit C Then Drink With Vit C | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 9 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Mean (Full Range); unit: years]
  years | 6.3 [6.0 to 6.6] | 6.4 [6.2 to 6.6] | 6.3 [6.0 to 6.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Philippines | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Iron Absorption
Description: Percentage of iron available for absorption from fortified oat drink with and without added vitamin C
Time Frame: 14 days after administration
Population: Per protocol
Measure: Mean (Standard Error); unit: percentage of Iron absorbed
Arm/Group | Fortified Oat Drink With Vitamin C | Fortified Oat Drink Without Vitamin C
Number analyzed (Participants) | 19 | 19
percentage of Iron absorbed | 7.14 (0.90) | 5.65 (0.54)

ADVERSE EVENTS:
Arm/Group | Drink With Vit C Then Drink Without Vit C | Drink Without Vitamin C Then Drink With Vit C
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
One of the isotopes was not detected in blood sample of 1 participant, therefore data from this participant was excluded from final per protocol analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 18 months from the time submitted to the sponsor for review.